CLINICAL TRIAL: NCT01278693
Title: Study of Treatment of Dyslipidemia for Hemodialysis
Brief Title: Effect of Oral L-carnitine Supplement on Lipid Profile, Anemia, and Quality of Life of Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASD-1213-11
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-08

CONDITIONS: Complication of Hemodialysis
Keywords: Renal failure, hemodialysis, dyslipidemia, L-carnitine.
MeSH Terms: conditions — Renal Insufficiency; Dyslipidemias | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Other): it is as like as L-carnitine in shape
  Interventions: Drug: placebo
- L-carnitine (Other): it is kind of supplement
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — 500 mg,twice daily, 16 weeks
  Arms: L-carnitine
Drug: placebo — 500 mg,twice daily, 16 weeks.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine Effect of oral L-carnitine supplement on lipid profile, anemia, and quality of life.

DETAILED DESCRIPTION:
In patients under maintenance hemodialysis several factors reduce the body stored carnitine which in turn affected dyslipidemia, anemia, and general health in these patients. The investigators evaluated the effect of oral L-carnitine supplementation on lipid profiles, anemia, and quality of life in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

being in the age range of 18-75 having the history of at least 12 weeks of hemodialysis and at least three times a week and each session almost for four hours having serum triglyceride or total cholesterol concentration >200 mg/dl or serum HDL concentration >40 mg/dl in the beginning of the study.

Exclusion Criteria:

taking carnitine supplement or the drug that interact with carnation lowering the seizure threshold in the last month being affected by liver function abnormalities, hypothyroidism, chronic infectious diseases (such as hepatitis), inflammatory diseases, CNS mass having the history of seizure.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
lipid profile | at sixteen weeks after admission

SECONDARY OUTCOMES:
anemia | at sixteen weeks after admission
quality of life | at sixteen weeks after admission

CONTACTS AND LOCATIONS:
Overall Officials: Mahnaz Moradi, MD, Study Chair — MD,research comittee
Locations (1):
- Noor university hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Derived] Nishioka N, Luo Y, Taniguchi T, Ohnishi T, Kimachi M, Ng RC, Watanabe N. Carnitine supplements for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013601. doi: 10.1002/14651858.CD013601.pub2. PMID 36472884